CLINICAL TRIAL: NCT00004842
Title: Pilot Study of Budesonide for Patients With Primary Sclerosing Cholangitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 199/13922; MAYOC-41296 (Other: Mayo Clinic); R03DK052344 (NIH)
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cholangitis, Sclerosing; Liver Cirrhosis, Biliary
Keywords: cirrhosis; gastrointestinal disorders; primary biliary cirrhosis; primary sclerosing cholangitis; rare disease
MeSH Terms: conditions — Cholangitis, Sclerosing; Liver Cirrhosis, Biliary; Fibrosis; Gastrointestinal Diseases; Rare Diseases | interventions — Budesonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Budesonide (Experimental): Oral budesonide
  Interventions: Drug: budesonide

INTERVENTIONS:
Drug: budesonide — Oral budesonide, 9 mg daily was administered for 1 year

SUMMARY:
OBJECTIVES: I. Assess the safety and effectiveness of budesonide in patients with primary sclerosing cholangitis or primary biliary cirrhosis experiencing a suboptimal response to ursodeoxycholic acid.

II. Estimate the efficacy of this therapy in these patient groups as a means of evaluating the feasibility of a long-term randomized trial.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive budesonide by mouth 3 times daily for a minimum of 6 months. If liver biochemistries become normal, dosage is reduced to once daily. Treatment discontinues after 1 year.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Pathologically confirmed primary sclerosing cholangitis (PSC) meeting the following criteria:

* Chronic cholestatic disease for at least 6 months
* Liver biopsy within the past 6 months compatible with the diagnosis of PSC Intra and/or extrahepatic biliary duct obstruction, beading, or narrowing

OR

Pathologically confirmed primary biliary cirrhosis (PBC) that is experiencing suboptimal response to ursodeoxycholic acid and meeting the following criteria:

* Chronic cholestatic liver disease for at least 6 months
* Positive antimitochondrial antibody
* No biliary obstruction by ultrasound, CT, or cholangiography
* Prior liver biopsy compatible with diagnosis of PBC
* Received ursodeoxycholic acid for at least 6 months

--Prior/Concurrent Therapy--

Biologic therapy:

* At least 3 months since prior D-penicillamine
* No planned transplantation for at least 1 year

Chemotherapy:

* At least 3 months (6 months for PBC) since prior cyclosporin, colchicine, azathioprine, or methotrexate
* At least 6 months since prior chlorambucil (PBC only)

Endocrine therapy: At least 3 months (6 months for PBC) since prior corticosteroids

Surgery: No prior intraductal stones or operations on the biliary tree except cholecystectomy (PSC only)

Other:

* At least 3 months since prior pentoxifylline, ursodeoxycholic acid, or nicotine (PSC only)
* At least 6 months since prior chenodeoxycholic acid (PBC only)

--Patient Characteristics--

Life expectancy: At least 3 years

Hematopoietic: Not specified

Hepatic:

* Alkaline phosphatase at least 2 times upper limits of normal
* No chronic hepatitis B infection
* No hepatitis C infection
* No autoimmune hepatitis
* Bilirubin no greater than 4 mg/dL (PBC only)

Cardiovascular: No severe cardiopulmonary disease

Other:

* No concurrent advanced malignancy
* At least 3 months since prior inflammatory bowel disease requiring specific treatment except maintenance therapy (PSC only)
* No anticipated need for transplantation within 1 year
* Not pregnant
* No liver disease of other etiology such as:

Chronic alcoholic liver disease

Hemochromatosis

Wilson's disease

Congenital biliary disease

Cholangiocarcinoma

No recurrent ascending cholangitis requiring hospitalization more than 2 times per year (PSC only)

At least 1 year since prior active peptic ulcer

No recurrent variceal bleeds

No spontaneous encephalopathy

No diuretic-resistant ascites

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 1997-05 (Actual); Primary Completion 1999-04 (Actual); Study Completion 1999-04 (Actual)

PRIMARY OUTCOMES:
Change in serum alkaline phosphatase | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Keith D. Lindor, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Angulo P, Jorgensen RA, Keach JC, Dickson ER, Smith C, Lindor KD. Oral budesonide in the treatment of patients with primary biliary cirrhosis with a suboptimal response to ursodeoxycholic acid. Hepatology. 2000 Feb;31(2):318-23. doi: 10.1002/hep.510310209. PMID 10655252